CLINICAL TRIAL: NCT00710541
Title: Non-invasive Ventilation in Patients With Severe Chronic Obstructive Pulmonary Disease and Lung Emphysema (COPD)
Brief Title: Non-invasive Ventilation in Severe Chronic Obstructive Pulmonary Disease(COPD)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The publication of a national guideline on NPPV precluded further recruitment.
Sponsor: Deutsche Lungenstiftung e.V. (Other)
Responsible Party: Principal Investigator, Dr. Thomas Koehnlein, M.D., Deutsche Lungenstiftung e.V.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COPD-Study; COPD1 (Other: Deutsche Lungenstiftung)
Record Dates: First submitted 2008-01-22; First posted 2008-07-04 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Chronic Obstructive Pulmonary Disease; Hypercapnia
Keywords: non invasive ventilation; COPD; hypercapnia; GOLD stage IV
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypercapnia | interventions — Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NPPV group (Experimental): Subjects in this arm receive standard COPD treatment, LTOT if indicated, and NPPV with ventilators designed for 'non invasive ventilation'(Resmed VPAP III ST-A, Weinmann Ventimotion, Tyco Healthcare Knight Star 330)
  Interventions: Device: ventilators designed for non invasive ventilation
- control gorup (No Intervention): Subjects in this arm receive standard COPD treatment and LTOT if indicated.

INTERVENTIONS:
Device: ventilators designed for non invasive ventilation — Patients are advised to use the ventilator for non invasive ventilation as long term treatment for at least 6 hours per day over one year.
  Other Names: Resmed VPAP III ST-A; Weinmann Ventimotion; Tyco Healthcare Knight Star 330
  Arms: NPPV group

SUMMARY:
Non-invasive ventilation is frequently applied in patients with acute exacerbation of COPD, but no evidence exists about the effect of long term application/home application.

This study tests the hypothesis, that a daily, 6 hour application of non-invasive ventilation over one year improves survival, exercise capacity, and quality of life in patients with advanced stages of COPD.

DETAILED DESCRIPTION:
The key problem of COPD (Chronic Obstructive Pulmonary Disease) is chronic inflammation and obstruction of the small airways. This results in a largely elevated flow resistance and work of breathing. The lungs develop enlarged air spaces (emphysema) with a reduction of alveoli and respiratory surface. Consequences are flattening of the diaphragm and alterations in the thoracic skeleton. COPD patients in advanced stages develop insufficiency of the muscular ventilatory pump. The ventilatory pump may decompensate, if the load of the muscles overruns their capacities. Besides that, an unphysiologically high proportion of the cardiac pump volume must be spent for the demands of the ventilatory muscles. Hypercapnia, and later hypoxaemia, are indicators of a decompensated ventilatory pump.

Theoretically, non-invasive ventilation (NIV) could be a treatment option for patients with advanced COPD and insufficiency of their ventilatory pump. Mechanical non-invasive ventilation provides support for the ventilatory muscles and might counterbalance the elevated intrinsic PEEP.

The physiologic and quality of life aspects of long term application on non-invasive ventilation (over at least one year) will be assessed in this study.

ELIGIBILITY:
Inclusion Criteria:

* Moderate or severe COPD with insufficiency of the ventilatory pump (according to GOLD stage IV). Stable disease since four weeks or more prior to randomisation. The COPD might be caused by whatever reason (smoking, Alpha-1 antitrypsin deficiency, ....). Smokers can be included.
* Capillary PCO2 of 7 kPa (51,8 mmHg) or maximally 10 kPa (74 mmHg), combined with a pH of 7.35 or above. These gases must be measured after 30 minutes breathing room air in sitting position. Patients on long term oxygen treatment must inhale oxygen in their prescribed dose.
* Only patients in the age of 18 years or above can be included.
* Written information about all aspects of the study (available in German language) must be provided for each patient. Written informed consent prior to any measure of this protocol is necessary for inclusion.

Exclusion Criteria:

* Patients with a PCO2 of 10 kPa (74 mmHg) or above. These patients can be re-evaluated for inclusion after 4 weeks.
* Diseases of the lung or thorax besides COPD: Advanced pulmonary fibrosis, advanced bronchiectases, active tuberculosis, post tuberculosis syndrome, pneumonia, severe kyphoscoliosis, tracheostoma, neuromuscular diseases, or any other disorder, which might result in elevated PCO2.
* Patients on NIV.
* Body mass index of 35 kg/m² or above.
* Severe cardiac disease, NYHA IV, instable angina, severe cardiac arrhythmia, especially of ventricular origin (atrial fibrillation is not an exclusion criterion).
* Malignoma
* Disorders of the basal brain nerves with derangement of swallowing, or reflexes of swallowing and choking.
* Local derangement of the face, skin, tongue, upper airways, larynx and upper oesophagus.
* Severe chronic diseases except COPD, hindering the patient to follow the schedule of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2004-10; Primary Completion 2011-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
all-cause mortality | one year

SECONDARY OUTCOMES:
exercise capacity | one year

CONTACTS AND LOCATIONS:
Overall Officials: Carl P Criée, Professor, Study Chair — Krankenhaus Göttingen-Weende, Klinik Lenglern
Locations (1):
- Medizinische Hochschule Hannover, Hanover, Germany

REFERENCES:
- [Background] Kohnlein T, Criee CP, Kohler D, Welte T, Laier-Groeneveld G. [Multicenter study on "non-invasive ventilation in patients with severe chronic obstructive pulmonary disease and emphysema(COPD)"]. Pneumologie. 2004 Aug;58(8):566-9. doi: 10.1055/s-2004-818542. German. PMID 15293170
- [Derived] Kohnlein T, Windisch W, Kohler D, Drabik A, Geiseler J, Hartl S, Karg O, Laier-Groeneveld G, Nava S, Schonhofer B, Schucher B, Wegscheider K, Criee CP, Welte T. Non-invasive positive pressure ventilation for the treatment of severe stable chronic obstructive pulmonary disease: a prospective, multicentre, randomised, controlled clinical trial. Lancet Respir Med. 2014 Sep;2(9):698-705. doi: 10.1016/S2213-2600(14)70153-5. Epub 2014 Jul 24. PMID 25066329